CLINICAL TRIAL: NCT06527755
Title: A Phase 1, Open-Label Study to Assess the Pharmacokinetics (PK), Pharmacodynamics (PD), Safety and Tolerability of Eplontersen Following Subcutaneous Administration of a Single Dose in Healthy Chinese Volunteers
Brief Title: A Study to Assess the PK, PD, Safety and Tolerability of Eplontersen in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D8450C00006
Record Dates: First submitted 2024-07-09; First posted 2024-07-30 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Transthyretin-mediated Amyloidosis
Keywords: Eplontersen; PK; PD; Safety; Tolerability; Open Label; Single Dose
MeSH Terms: interventions — Injections; eplontersen

STUDY DESIGN:
Intervention Model Description: This study is a single-arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eplontersen (Experimental): Single arm
  Interventions: Drug: Eplontersen Solution for Injection

INTERVENTIONS:
Drug: Eplontersen Solution for Injection — an autoinjector with 0.8 mL deliverable volume (at 56 mg/mL concentration) will be provided, total dose is 45 mg.
  Other Names: Eplontersen

SUMMARY:
This is a Phase 1 study to assess the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of eplontersen following single dosing in healthy Chinese participants. The objectives of the study are: to characterize the pharmacokinetic (PK) profiles and the pharmacodynamic (PD) profiles, and to evaluate the safety and tolerability and the immunogenicity of eplontersen following subcutaneous administration of a single 45 mg dose in healthy Chinese participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-dose, single-arm study to assess the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of eplontersen following subcutaneous (SC) administration in healthy Chinese male and female participants. Approximately 12 healthy Chinese participants, aged 18 to 60 years, will be assigned to study intervention of a signle dose of eplontersen 45 mg following subcutaneous administration. Including the administration dosing day, the follow-up period is total of 92 days. The primary objective of this study is to characterize the PK profile of eplontersen, the PK parameters for eplontersen including, but not limited to: Cmax, tmax, t½λz, AUC0-24h, and AUC0-168h. The secondary objective of this study is to characterize the PD profiles of eplontersen, this includes the measures of change and percent change from baseline in serum TTR levels at specified timepoints. The safety objective of this study is to evaluate the safety and tolerability of eplontersen, this includes the measures of AEs/SAEs, vital signs, physical examinations, safety laboratory assessments and 12-lead ECG. Also the exploratory objective of this study is to evaluate the immunogenicity of eplontersen, this includes the measures of but not limited to anti-drug antibodies (ADA) prevalence and incidence, different ADA status at specified timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements.
2. Healthy* Chinese males or females of non-childbearing potential, aged 18 to 60 inclusive at the time of informed consent.

   *Participants will be confirmed to be healthy according to the medical history, electrocardiogram (ECG), vital signs, laboratory results, and physical examination as determined by the Investigator.
3. Females must be non-pregnant and non-lactating, and either surgically sterile (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea without an alternative medical cause and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory involved. Males must be surgically sterile or abstinent*, or if engaged in sexual relations with a female of child-bearing potential, the participant must be using an highly effective contraceptive method from the time of signing the informed consent form until at least 24 weeks after study intervention administration.

   * Abstinence is only acceptable as true abstinence, ie, when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a study and withdrawal are not acceptable methods of contraception.
4. Willing to refrain from strenuous exercise/activity (eg, heavy lifting, weight training, intense aerobics classes) for at least 72 hours prior to study visits.
5. Weight ≥ 50 kg and body mass index (BMI) of 19 to 30 kg/m2 at screening (including cutoff).

   BMI = weight (kg)/height2 (m2).
6. Willingness to take vitamin A supplements (recommended daily allowance [RDA] of approximately 3000 IU/day until the last post-treatment follow-up visit [Day 92; 13 weeks after the dosing]).

Exclusion Criteria:

1. Clinically significant abnormalities in medical history (eg, major surgery within 6 months of screening, history or presence of hepatic, renal, hematological, endocrine, or cardiovascular disease) or physical examination.
2. Screening laboratory results as follows, or any other clinically significant abnormalities in screening laboratory values that would render a participant unsuitable for inclusion:

   * Random spot urine protein/creatinine ratio (UPCR) ≥ 200 mg/g. In the event of UPCR above this threshold ineligibility may be confirmed by a repeat random spot UPCR ≥ 200 mg/g or a 24-hour urine protein ≥ 200 mg/24 hour;
   * Positive test for blood (including trace) on urinalysis that is subsequently confirmed with urine microscopy showing > 5 red blood cells per high power field;
   * Alanine transaminase (ALT), aspartate aminotransferase (AST), bilirubin, alkaline phosphatase (ALP), serum creatinine, and blood urea > upper limit of normal (ULN);
   * Fasting blood glucose > ULN;
   * Platelet count < lower limit of normal (LLN);
   * Estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) ≤ 60 mL/min/1.73m2.
3. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Day 1.
4. Unwillingness to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator.
5. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis B antigen, and hepatitis C antibody.
6. Uncontrolled hypertension (systolic blood pressure [BP] > 160 mmHg, or diastolic BP > 100 mmHg).
7. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
8. Treatment with another investigational drug, biological agent, or device within 1 month of screening, or 5 half-lives of study intervention, whichever is longer.
9. Previous treatment with an oligonucleotide (including small interfering ribonucleic acid) within 4 months of screening if single dose received, or within 12 months of screening if multiple doses received (exception for SARS-Cov2 vaccines [both mRNA and viral vector vaccines]; any vaccine should be administered at least 7 days prior to study intervention).
10. History of bleeding diathesis or coagulopathy.
11. Regular use of alcohol within 6 months prior to screening (> 7 drinks/wk for females, > 14 drinks/wk for males [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor]), or use of soft drugs (such as marijuana) within 3 months prior to screening, or hard drugs (such as cocaine and phencyclidine) within 1 year prior to screening, or positive urine drug and alcohol screen at screening.
12. Concomitant medication restrictions including any prescription and over-the-counter (OTC) and herbal remedies, other than occasional acetaminophen (paracetamol) or ibuprofen unless authorized by the Study Clinical Lead.
13. Smoking limitations: smoking > 10 cigarettes a day.
14. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening.
15. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the participant unsuitable for inclusion, or could interfere with the participant participating in or completing the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
PK parameters: Maximum Observed Concentration(Cmax) | collect PK sample in pre-dose of Day 1 and 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours of post-dose, and in Day 8, Day 15, Day 29, Day 50, Day 71, Day 92
  To characterize the pharmacokinetic (PK) profiles of eplontersen following subcutaneous administration of a single 45 mg dose in healthy Chinese participants
PK parameters: Time to Maximal Concentration (tmax) | collect PK sample in pre-dose of Day 1 and 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours of post-dose, and in Day 8, Day 15, Day 29, Day 50, Day 71, Day 92
  To characterize the pharmacokinetic (PK) profiles of eplontersen following subcutaneous administration of a single 45 mg dose in healthy Chinese participants
PK parameters: Plasma Half-life Associated with the Apparent Terminal Elimination Phase (t½λz) | collect PK sample in pre-dose of Day 1 and 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours of post-dose, and in Day 8, Day 15, Day 29, Day 50, Day 71, Day 92
  To characterize the pharmacokinetic (PK) profiles of eplontersen following subcutaneous administration of a single 45 mg dose in healthy Chinese participants
PK parameters: Area Under Plasma Concentration-time Curve (0-24 hours) (AUC0-24h) | collect PK sample in pre-dose of Day 1 and 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours of post-dose, and in Day 8, Day 15, Day 29, Day 50, Day 71, Day 92
  To characterize the pharmacokinetic (PK) profiles of eplontersen following subcutaneous administration of a single 45 mg dose in healthy Chinese participants
PK parameters: Area Under Plasma Concentration-time Curve (0-168 hours) (AUC0-168h) | collect PK sample in pre-dose of Day 1 and 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours of post-dose, and in Day 8, Day 15, Day 29, Day 50, Day 71, Day 92
  To characterize the pharmacokinetic (PK) profiles of eplontersen following subcutaneous administration of a single 45 mg dose in healthy Chinese participants

SECONDARY OUTCOMES:
The change and percent change from baseline in serum (Transthyretin) TTR levels at specified timepoints | collect PD sample in screening visit, pre-dose of Day 1 and Day 8, Day 15, Day 29, Day 50, Day 71, Day 92
  To characterize the pharmacodynamic (PD) profiles of eplontersen following subcutaneous administration of a single 45 mg dose in healthy Chinese participant

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lin, Medical PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Research Site, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual subject-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://www.astrazenecaclinicaltrials.com/our-transparency-commitments/ AZ accept request for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at: https://www.astrazenecaclinicaltrials.com/our-transparency-commitments/.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statement at: https://www.astrazenecaclinicaltrials.com/our-transparency-commitments/.
URL: https://vivli.org/